CLINICAL TRIAL: NCT04057638
Title: Combined Craniomaxillofacial and Upper Extremity Allotransplantation
Brief Title: Craniomaxillofacial and Upper Extremity Allotransplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: s19-00621
Record Dates: First submitted 2019-08-06; First posted 2019-08-15 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Face Injuries; Hand Injuries; Craniofacial Injuries; Upper Extremity Injuries; Facial Injuries; Facial Deformity
Keywords: Transplants; Transplantation; Craniomaxillofacial Transplantation; Upper Extremity Transplantation; Vascularized Composite Allotransplantation (VCA)
MeSH Terms: conditions — Facial Injuries; Hand Injuries

STUDY DESIGN:
Intervention Model Description: This is a prospective longitudinal observational analysis of functional and aesthetic outcomes after treatment of severe facial defects and upper extremity injuries with microvascular composite tissue allotransplantation. There will only be the treatment group in this study, which undergoes microvascular VCA transplantation. There will be no randomization, placebo or control groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): There will only be the treatment group in this study, which undergoes microvascular VCA transplantation. There will be no randomization, placebo or control groups.
  Interventions: Procedure: Combined Craniomaxillofacial and Upper Extremity Allotransplantation

INTERVENTIONS:
Procedure: Combined Craniomaxillofacial and Upper Extremity Allotransplantation — Combined Craniomaxillofacial and Upper Extremity Allotransplantation

SUMMARY:
The purpose of this study is to evaluate functional and aesthetic outcomes of combined facial and upper extremity composite tissue allografts on patients who have not achieved functional and aesthetic outcomes with conventional reconstructive surgical strategies and prosthetic devices.

DETAILED DESCRIPTION:
The purpose of this study is to see if an investigational surgery that transfers tissue from a non-living donor to a living individual will help restore greater function, appearance, and sensation to the face and upper extremity areas of individuals who have suffered injury to those areas. Upper extremity constitutes the part of the body including arm, forearm and hand. This procedure is called combined craniomaxillofacial and upper extremity allotransplantation or "combined face and upper extremity transplant".

This study will also collect data on how patients do during and after having a combined face and upper extremity transplant from a nonliving donor. Recovery and outcomes will be observed through clinical exams, x-rays, blood and tissue tests, and other associated evaluations at all follow up visits.

Participants are invited to take part in this research study who have suffered severe injury to the face and upper extremity and previous surgeries to repair the injury have not restored function, appearance, and sensation. Participants must have attempted a trial of prosthetics (artificial upper extremity), if at all possible.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated all required Institutional Review Board (IRB) approved consent forms.
* Male or female recipient between the ages of 18-64 years. Recipients do not need to be of the same sex as the donor.
* Facial composite tissue defect requiring facial transplantation as determined by the treating Plastic and Reconstructive Surgeon. Inclusive facial functional subunit tissue loss. Including but not limited to irreparable peri-oral, peri-orbital, and peri-nasal damage.
* Missing part of one or both hands and forearms.
* Must be HIV negative at the time of transplant.
* Crossmatch is negative at the time of transplant.
* Patient has been encouraged to seek a second opinion from a Plastic Surgeon with specialized focus in facial reconstruction.
* Patient has been encouraged to seek a second opinion from a Plastic Surgeon with specialized focus in upper extremity reconstruction.
* Willingness to participate in ongoing psychiatric, psychological and social work evaluations prior to and post-transplant surgery.
* The subject is able to complete pre-transplant examination and screening procedures.
* Patient has been approved by Patient Selection Committee for placement on the recipient waiting list.
* The subject is willing to continue immunosuppression regimen as directed by treating physician.
* Subject is willing and able to return to follow-up visits as described in treatment plan.
* Subjects must have autogenous tissue options available for reconstruction in event of graft failure.
* Normal glomerular filtration rate (GFR) >60.
* Negative pregnancy test within 48hrs of transplant for women of childbearing age and who agree to use a reliable form of contraception for one year following transplant.

Exclusion Criteria:

* Uncontrolled infection or severe concomitant diseases which would exclude the recipient from transplantation
* Serious co-morbidities
* Positive serology for HIV; Hepatitis B Antigen
* Active malignancy within 5 years with the exclusion of non-melanoma
* Substance abuse disorders not currently under control (as determined by the Michigan Alcohol Screening Test - see Appendix N.1: Subjects with a score of 3 or more will be excluded)
* Body Dysmorphic disorder (see Appendix N.2 for screening tool). Less severe psychiatric conditions are addressed on a case by case basis
* Active Severe Psychiatric Illness
* Cognitive limitations affecting the patient's ability to provide informed consent
* Recent history of medical non-adherence
* Unstable social situation as evidence by lack of stable housing and/or lack of a supportive significant other.
* Recent history of medical non-adherence.
* Lack of stable housing and/or supportive significant other/caregiver throughout all phases of the study
* Currently active smoker within 1 year
* Subjects with any cognitive deficits related to a traumatic brain injury (TBI) and or any organic neurological disorders
* Any other psychological status that would hinder the success or safety of the transplantation.
* Level of amputation proximal to mid-humerus: some presence of proximal muscles is required to motor a functioning hand.
* Congenital Abnormalities: co-existent absence/atrophy/agenesis of any tissue may affect post-transplant results
* History of amputation of less than six months: subject must be allowed to attempt prosthetic use prior to hand transplantation. This can be waived in cases where the recipient requires amputation/revision of the transplant site at the time of transplantation. However, if at all possible, it is highly encouraged that the patient has ruled out prosthetics as an alternative to transplantation.
* Blindness: blind amputees may be poor candidates because sensory return in the hand may not provide sufficient protective sensation
* Pregnancy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-06-17 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in function of the transplanted facial segment | Monthly for 6 months, every 6 months for 2 years, then annually up to year 5
  This will be measured using electromyogram (EMG)
Change in function of the transplanted facial segment | Monthly for 6 months, every 6 months for 2 years, then annually up to year 5
  This will be measured using nerve conduction studies (NCS)
Change in function of the transplanted facial segment | Monthly for 6 months, every 6 months for 2 years, then annually up to year 5
  This will be measured using computerized tomography angiogram (CTA)
Change in function of the transplanted facial segment | Monthly for 6 months, every 6 months for 2 years, then annually up to year 5
  This will be measured using magnetic resonance imaging (MRI)
Change in function of the transplanted facial segment | Monthly for 6 months, every 6 months for 2 years, then annually up to year 5
  This will be measured using vision exams
Change in function of the upper extremity transplant | Monthly for 6 months, every 6 months for 2 years, then annually up to year 5
  This will be measured using pathology samples to check for rejection
Change in function of the upper extremity transplant | Monthly for 6 months, every 6 months for 2 years, then annually up to year 5
  This will be measured using electromyogram (EMG)
Change in function of the upper extremity transplant | Monthly for 6 months, every 6 months for 2 years, then annually up to year 5
  This will be measured using nerve conduction studies (NCS)
Change in function of the upper extremity transplant | Monthly for 6 months, every 6 months for 2 years, then annually up to year 5
  This will be measured using computerized tomography angiogram (CTA)
Change in function of the upper extremity transplant | Monthly for 6 months, every 6 months for 2 years, then annually up to year 5
  This will be measured using magnetic resonance imaging (MRI)
Change in appearance of the transplanted facial segment | Monthly for 6 months, every 6 months for 2 years, then annually up to year 5
  This will be measured using photography
Change in appearance of the upper extremity transplant | Monthly for 6 months, every 6 months for 2 years, then annually up to year 5
  This will be measured using photography

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Rodriguez, MD, DDS, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States